CLINICAL TRIAL: NCT06320171
Title: Efectivity of Non-invasive Neuromodulation in Parasympathic Nervous System and Vascular System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Vanesa Abuín, Associated Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 240118,2024-481
Record Dates: First submitted 2024-02-22; First posted 2024-03-20 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The intervention in the study involves a unique application of 20min of NESA microcurrents
  During the intervention, patients were seated comfortably on a sofa with their backs supported. NESA, a portable, noninvasive neuromodulation device, delivered low-frequency (1.3-14.28 Hz), low-intensity (0.1-0.9 mA), low-voltage (±3 V) microcurrents through 24 electrodes placed on the distal nerve endings of the wrists and ankles (six electrodes per limb). Direct stimulation of the autonomic nervous system was achieved using program 7 of the device with a directional electrode placed at the level of the C7 spinous process. This configuration established a circulating bioelectric circuit within the body, stimulating the autonomic nervous system below the patient's sensory threshold
  Interventions: Device: Non-Invasive neuromodulation
- Placebo (Placebo Comparator): The placebo group followed the same procedure, except that no current was applied during their 20-minute session.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Non-Invasive neuromodulation — Direct stimulation of the autonomic nervous system was achieved using Program 7 (P7) of the device, with a directional electrode positioned at the level of the C7 spinous process. P7 delivered a biphasic polarity current with oscillatory frequencies ranging from 1.92 to 14.29 Hz and variable intensities between 0.1 and 0.9 mA.
  Arms: Experimental
Other: Placebo — The placebo group followed the same procedure, except that no current was applied during their 20-minute session.
  Arms: Placebo

SUMMARY:
The aim of the present study is to evaluate the acute effect immediately after the application of the NESA treatment in healthy participants in vascular sonographic variables measured in the left CCA such as the LD, IMT and PSV, as well as systolic (sBP) and diastolic blood (dBP) pressure and heart rate (HR). The investigators hypothesized that NESA application will induce a direct influence in the vascular tone through the stimulation of the ANS and the parasympathetic nerve system. This premise is based on the fact that non-invasive NESA neuromodulation enhance the autonomic regulation of vascular tone and endothelial function.

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the acute effect immediately after the application of the NESA treatment in healthy participants in vascular sonographic variables measured in the left CCA such as the LD, IMT and PSV, as well as systolic (sBP) and diastolic blood (dBP) pressure and heart rate (HR). We hypothesize that NESA application will induce a direct influence in the vascular tone through the stimulation of the ANS and the parasympathetic nerve system. This premise is based on the fact that non-invasive NESA neuromodulation enhance the autonomic regulation of vascular tone and endothelial function.A total sample of forty participants (N = 40; mean age 26.6 ± 6.7 years) were recruited for participation in the study. Prior to entering the study, all participants received information about the study and signed a consent form to participate. The study subjects were divided into two equally distributed groups (A: NESA = 20; B: Placebo = 20) and were blinded to the study group allocation. Participants in the placebo group underwent the same procedural phases as those in the intervention group. However, for the placebo group, the device was set to deliver a low-intensity current below the sensory threshold, effectively rendering it inactive from the participants' perspective.

ELIGIBILITY:
Inclusion:

- Age between: 18-55 years, both sexes.

Exclusion:

* Cardiovascular disease.
* Specific pharmacology.
* Hypertension.
* Diabetes.
* Systemic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic Blood Pressure: | before the intervention, and 10 minutes after the intervention
  The pressure in the arteries during the contraction of the heart muscle. Measured with sphingomanometer.
Heart rate | Before the intervention, and 10 minutes after the intervention
  Hearbears per minute

SECONDARY OUTCOMES:
Ultrasonographic variables: Cross-sectional area of the jugular vein | Before the intervention, and 10 minutes after the intervention
  Cross-sectional area of the jugular vein
Ultrasonographic variables:Cross-sectional area of the common carotid | Before the intervention, and 10 minutes after the intervention
  Cross-sectional area of the common carotid
Ultrasonographic variables:Thickness of the common carotid | Before the intervention, and 10 minutes after the intervention
  Thickness of the common carotid
Ultrasonographic variables:Peak systolic velocity. | Before the intervention, and 10 minutes after the intervention
  Peak systolic velocity.
Cortisol measurement | Before the intervention, and 10 minutes after the intervention
  Measure of cortisol level.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrod, Villaviciosa de Odón, Spain

IPD SHARING:
Plan to Share IPD: No